CLINICAL TRIAL: NCT03623191
Title: Clinical Aspect of Erosive Pustular Dermatosis of the Leg
Acronym: Clin-EPDL
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2017Ao006
Record Dates: First submitted 2018-08-07; First posted 2018-08-09 (Actual); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Erosive Pustular Dermatosis of the Leg
Keywords: Erosive pustular dermatosis of the leg; Erosive pustular dermatosis of the scalp; Venous insufficiency
MeSH Terms: conditions — Venous Insufficiency | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with erosive pustular dermatosis of the leg
  Interventions: Other: Clinical examination

INTERVENTIONS:
Other: Clinical examination

SUMMARY:
Erosive pustular dermatosis of the leg is a fairlyrecent clinical entity that was described the first time in 1987.

Diagnosis of erosive pustular dermatosis of the leg is made on clinical grounds. It presents as non-follicular pustules of variable size and numbers that rapidly give way to erosions and crusts on one or both legs, and which are found in particular on the anterior aspect of the middle third of the leg (. The lesions are of chronic progression, despite topical therapy. Erosive pustular dermatosis of the leg is seen in elderly patients, mainly female, and may be associated with chronic venous insufficiency or cutaneous atrophy. In the absence of specific criteria and because of the existence of misleading clinical forms, diagnosis is based upon exclusion.

DETAILED DESCRIPTION:
The primary objective of this investigation was to describe the different clinical aspects of cases of Erosive pustular dermatosis of the leg.

ELIGIBILITY:
Inclusion Criteria:

- non-follicular pustules and multiple erosions on one or both legs showing no evidence of improvement after application of compression in the event of clinical signs of chronic venous insufficiency and showing no improvement following treatment with local and/or systemic antibacterial therapy, fungal samples from the pustules negative on direct examination, negative direct immunofluorescence results for biopsy samples (taken from around the lesion)

Exclusion Criteria:

- age < 18 years old

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with erosive pustular dermatosis of the leg
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2014-10-01 (Actual); Study Completion 2015-06-01 (Actual)

PRIMARY OUTCOMES:
Lesions location | Day 0
  Anterior or posterior leg face
number of lesions | Day 0
  Less than 10 erosions, between 10 and 50 erosions and more than 50 erosions
Presence of chronic venous insufficiency | Day 0
  Diagnosis based on the CEAP 2004 Score (Eklöf B, Rutherford RB, Bergan JJ, Carpentier PH, GloviczkiP, Kistner RL, et al. Revision of the CEAP classification forchronic venous disorders: consensus statement. J Vasc Surg2004;40:1248-52)

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France

REFERENCES:
- [Background] Nicol P, Perceau G, Barbe C, Bernard P; members of GAD. Erosive pustular dermatosis of the leg: A prospective, multicentre, observational study of 36 cases. Ann Dermatol Venereol. 2017 Oct;144(10):582-588. doi: 10.1016/j.annder.2017.02.007. Epub 2017 May 19. PMID 28532589